CLINICAL TRIAL: NCT05110209
Title: Real-world Evaluation of Prevalence of Ocular Adverse Events in Patients With Neovascular (Wet) Agerelated Macular Degeneration (AMD) Who Received Anti-VEGF Agents (IRIS Registry)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AUS20
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept; Ranibizumab; Bevacizumab; Off-Label Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aflibercept: Patients/patient eyes who were treated only with aflibercept in 2019
  Interventions: Other: Aflibercept
- Ranibizumab: Patients/patient eyes who were treated only with ranibizumab in 2019
  Interventions: Other: Ranibizumab
- Bevacizumab: Patients/patient eyes who were treated only with bevacizumab in 2019
  Interventions: Other: Bevacizumab
- ≥2 Different Anti- VEFGFs: Patients/patient eyes who were treated with ≥2 different anti-VEGFs in 2019

INTERVENTIONS:
Other: Aflibercept — intravitreal injection
  Other Names: EYLEA®
  Groups: Aflibercept
Other: Ranibizumab — intravitreal injection
  Other Names: LUCENTIS®
  Groups: Ranibizumab
Other: Bevacizumab — intravitreal injection
  Other Names: AVASTIN®; off-label use
  Groups: Bevacizumab

SUMMARY:
In this cross-sectional study of patients with wet AMD who received ≥1 anti-VEGF injection (excluding brolucizumab), evidence was generated to describe the period prevalence of specific ocular AEs. The study was conducted using the IRIS Registry, and all results were based on the study period from 01/01/2019 to 12/31/2019.

DETAILED DESCRIPTION:
This was a retrospective cohort study of eyes in adult patients with a diagnosis of wet AMD who were treated with anti-VEGF agents from 01/01/2019 to 12/31/2019.

IRIS Registry data from 01/01/2019 to 12/31/2019 for patients with a diagnosis of wet AMD who were treated with ≥1 anti-VEGF agent (excluding brolucizumab) were included.

* Identification period: Patients fulfilling the selection criteria during the period from 01/01/2019 to 12/31/2019 were identified
* Index date: 01/01/2019
* Study Period: 01/01/2019 to 12/31/2019
* Pre-index period: 01/01/2018 to 12/31/2018
* Post-index period: 01/01/2019 to 12/31/2019

ELIGIBILITY:
Inclusion Criteria:

* ≥1 International Classification of Diseases, Clinical Modification-9/10 CM (ICD- 9/10) code for wet AMD in 2019
* ≥1 Healthcare Common Procedure Coding System (HCPCS) code (J code) or National Drug Code (NDC) code for treatment with an anti-VEGF agent (excluding brolucizumab) in 2019
* ≥18 years old in 2019
* ≥2 wet AMD-related office visits in 2019

Exclusion Criteria:

* Patient eyes that received >1 type of anti-VEGF treatment on the same date
* Patient eyes that did not have laterality any time during 2018-2019
* Treatment with brolucizumab during 2019

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IRIS Registry data from 01/01/2019 to 12/31/2019 for patients with a diagnosis of wet AMD who were treated with ≥1 anti-VEGF agent (excluding brolucizumab) were included.
Sampling Method: Probability Sample
Enrollment: 331541 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with Intraocular Inflammation (IOI) Adverse events (AEs) who were treated with anti-VEGF agents | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  Period prevalence of IOI in patients with wet AMD who were treated with anti- VEGF agents (excluding brolucizumab) over a one-year period in 2019 was assessed.

SECONDARY OUTCOMES:
Age | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  Age information was reported
Gender information | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  Gender information was reported
Number of patients at various Patient Region | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  Patient regions: Northeast, Midwest, South, West, Unknown
Number of patients with Insurance type | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  Private, Medicare, Medicare Advantage, Medicaid, Other
Number of patients with Laterality of wet Age-related macular degeneration (AMD) | Index date (defined as the date of first injection - 01/01/2019)
  Laterality of wet AMD: Unilateral, Bilateral
Number of patient eyes with the Provider specialty on date of first anti-VEGF injection | earliest claim of anti-VEGF injection over a one-year period from 01/012019 to 31/12/2019
  The following types were included: Retina specialist, General ophthalmologist
Number of patient eyes treated with anti-VEGF agent | Index date (defined as the date of first injection - 01/01/2019)
  The following types were included OD [eye, right], OS [eye, left], Unspecified
Number of anti-VEGF injections | over a one-year period from 01/012019 to 31/12/2019
  Anti-VEGF utilization in patients with wet AMD who were treated with anti- VEGF agents (excluding brolucizumab) over a one-year period was assessed. Measured at the patient level and patient-eye level.
Number of patients with other ocular AEs in patients with wet AMD who were treated with anti-VEGF agents (excluding brolucizumab) | over a one-year period from 01/012019 to 31/12/2019
  The following types were included:
  1. Key ocular AEs
  2. IOI events
  3. RVO events
  4. Unspecified RO
  5. Autoimmune disorders (systemic lupus erythematosus [SLE], Behcet's disease, sarcoidosis, VKH disease, HLA-B27 syndromes, Drug hypersensitivity)
  6. RV without RO (RAO and/or RVO)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CRTH258AUS20 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17877